CLINICAL TRIAL: NCT03732079
Title: The Correlation Between Inferior Vena Caval Diameter and the Volume of Postpartum Blood Loss
Brief Title: Inferior Vena Cava Diameter and Postpartum Hemorrhage
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Sponsor
Other Study IDs: HaEmek
Record Dates: First submitted 2018-11-04; First posted 2018-11-06 (Actual); Last update posted 2018-11-06 (Actual); Status verified 2018-11

CONDITIONS: Other Immediate Postpartum Hemorrhage, With Delivery
Keywords: Inferior Vena Cava Diameter
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- Research group: Women with early postpartum hemorrhage.
  Interventions: Diagnostic Test: Ultrasound
- Control group: Postpartum women without abnormal bleeding.
  Interventions: Diagnostic Test: Ultrasound

INTERVENTIONS:
Diagnostic Test: Ultrasound — Ultrasound to measure the IVC diameter. The IVC diameter will be measured in the inspirium and the expirium, and the collapsibility index will be recorded.

SUMMARY:
Excessive bleeding after normal birth or cesarean section is defined as blood loss of 1000 mL or more (clinically estimated) within 24 hours after birth. It occurs in about 5% among postpartum women. Postpartum hemorrhage is a leading cause of morbidity and mortality among women giving birth. Postpartum hemorrhage may lead to hemorrhagic shock, renal failure, respiratory failure, need for surgical intervention, blood transfusion and hysterectomy.

The cornerstone of effective treatment is rapid diagnosis and intervention in time. However, in a number of cases there is an underestimation of the volume of blood loss which may lead to delay in diagnosis and treatment. The consequences are even graver in women who delivered by a cesarean section, since unlike a normal birth in which the bleeding is external and visible, the bleeding is usually intra-abdominal, and so the delay in diagnosis may be even longer.

The Inferior Vena Cava (IVC) is a flexible blood vessel sensitive to intravascular blood volume, and its diameter varies accordingly. Its diameter reflects the pressure in the right atrium, which is a measure of the cardiac preload. A number of studies have shown that the IVC diameter changes, before the variations in vital and clinical signs.

Recently, IVC diameter has been assessed as an assessment of intravenous fluid balance in hemodynamically stable patients with a risk of sub-volume shock. The authors concluded that the IVC measurement is a good noninvasive method, compared to catheter insertion into the right atrium, and it is available as a bedside procedure.

In obstetrics the use of IVC to determine blood loos was not widely examined and there is no information regarding the use of IVC diameter as a predictor or as a detection method of postpartum bleeding.

In this study the investigators aim to examine the correlation between IVC diameter and the volume of postpartum blood loss.

ELIGIBILITY:
Inclusion Criteria:

* Women over the age of 18 after birth
* Single pregnancy
* Vaginal birth
* Term pregnancy (gestational age between week 37-42)
* The newborn is appropriate for gestational age (10-90 percentile)

Exclusion Criteria:

* Gestational or pre-pregnancy hypertension
* Heart, liver, or chronic kidney disease
* Women who delivered newborn with major malformation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — postpartum women
Study Population: Postpartum women.
Sampling Method: Probability Sample
Enrollment: 108 (Estimated)
Dates: Start 2018-11-10 (Estimated); Primary Completion 2019-04-30 (Estimated); Study Completion 2019-04-30 (Estimated)

PRIMARY OUTCOMES:
To examine the correlation between IVC diameter and the volume of postpartum blood loss. | 6 months

SECONDARY OUTCOMES:
To create a normogram of IVC diameter in postpartum women and to check whether there is a cutt-of value that appears before the onset of clinical signs of blood loss. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Manal Massalha, Massalha, Principal Investigator — Emek Medical Center

REFERENCES:
- [Result] Committee on Practice Bulletins-Obstetrics. Practice Bulletin No. 183: Postpartum Hemorrhage. Obstet Gynecol. 2017 Oct;130(4):e168-e186. doi: 10.1097/AOG.0000000000002351. PMID 28937571
- [Result] Callaghan WM, Kuklina EV, Berg CJ. Trends in postpartum hemorrhage: United States, 1994-2006. Am J Obstet Gynecol. 2010 Apr;202(4):353.e1-6. doi: 10.1016/j.ajog.2010.01.011. PMID 20350642
- [Result] Byeon K, Choi JO, Yang JH, Sung J, Park SW, Oh JK, Hong KP. The response of the vena cava to abdominal breathing. J Altern Complement Med. 2012 Feb;18(2):153-7. doi: 10.1089/acm.2010.0656. PMID 22339104
- [Result] Grant E, Rendano F, Sevinc E, Gammelgaard J, Holm HH, Gronvall S. Normal inferior vena cava: caliber changes observed by dynamic ultrasound. AJR Am J Roentgenol. 1980 Aug;135(2):335-8. doi: 10.2214/ajr.135.2.335. PMID 6773338
- [Result] Kusaba T, Yamaguchi K, Oda H, Harada T. Echography of inferior vena cava for estimating fluid removed from patients undergoing hemodialysis. Nihon Jinzo Gakkai Shi. 1994 Aug;36(8):914-20. PMID 7933667
- [Result] Lyon M, Blaivas M, Brannam L. Sonographic measurement of the inferior vena cava as a marker of blood loss. Am J Emerg Med. 2005 Jan;23(1):45-50. doi: 10.1016/j.ajem.2004.01.004. PMID 15672337
- [Result] Rahman NH, Ahmad R, Kareem MM, Mohammed MI. Ultrasonographic assessment of inferior vena cava/abdominal aorta diameter index: a new approach of assessing hypovolemic shock class 1. Int J Emerg Med. 2016 Dec;9(1):8. doi: 10.1186/s12245-016-0101-z. Epub 2016 Feb 19. PMID 26894896
- [Result] Hernandez CA, Reed KL, Juneman EB, Cohen WR. Changes in Sonographically Measured Inferior Vena Caval Diameter in Response to Fluid Loading in Term Pregnancy. J Ultrasound Med. 2016 Feb;35(2):389-94. doi: 10.7863/ultra.15.04036. Epub 2016 Jan 18. PMID 26782160
- [Result] Ryo E, Unno N, Hagino D, Kozuma S, Nagasaka T, Taketani Y. Inferior vena cava diameter and the risk of pregnancy-induced hypertension and fetal compromise. Int J Gynaecol Obstet. 1999 May;65(2):143-8. doi: 10.1016/s0020-7292(99)00027-2. PMID 10405058